CLINICAL TRIAL: NCT01168518
Title: Performance of the New Generation of Sorin Group Brady Leads In a Normal Hospital Practice
Brief Title: An Observational Study on the Sorin Group New Brady Leads XFine and Beflex
Acronym: XFine & Beflex
Status: Completed | Type: Observational
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: RLEA01-FINE; RLEA01
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Pacing Leads Implantation
Keywords: Evaluate the Sorin Group new passive- and active- fixation pacing leads

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study is a non-interventional multi-centre, prospective study.

The aim of the study is to evaluate the Sorin Group new passive- and active- fixation pacing leads. We plan to assess the acute and short term lead dislodgment rate (within the first three months following implantation) correlated with the type of lead (active- or passive- fixation). Further, we are collecting data related to leads handling and leads electrical performances

DETAILED DESCRIPTION:
The primary objective of this observational study is to assess the acute rate of dislodgment of the new Sorin group range of active- and passive- fixation leads up to 3 months following implant.

Assessment of electrical performances (pacing threshold, sensing amplitude, impedance) of the leads at implant and during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* The implanted lead must allow the measurement of pacing threshold at 0.5ms, R-wave or P-wave amplitude and impedance of the lead.
* Included patients may receive more than one lead under evaluation.

Exclusion Criteria:

* Any contraindication to endocavitary lead implantation;
* Inability to understand the purpose of the study or refusal to co-operate.
* Geographically unstable or unavailability for scheduled M1-M3 follow-up at the implanting centre as defined in the investigational plan.
* Patient of minor age (<18)
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient implanted with an endocavitary pacing lead (atrial and/or ventricular) connected to a single, double or triple chamber pacemaker or defibrillator.
Sampling Method: Probability Sample
Enrollment: 2254 (Actual)
Dates: Start 2008-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Lead dislodgment rate in acute phase | Lead dislodgment
  Ventricular active fixation leads = 1.57%; Ventricular passive fixation leads = 3.23%, Atrial active fixation leads = 1.04%

CONTACTS AND LOCATIONS:
Overall Officials: Henri Benkemoun, MD, Principal Investigator — Unité de Cardiologie et Rythmologie Interventionelle, Perpignan France
Locations (1):
- Clinique St Pierre, Perpignan, Perpignan, France